CLINICAL TRIAL: NCT01402518
Title: Observational Study of the Per-Oral Endoscopic Myotomy (POEM) Procedure
Brief Title: Per-Oral Endoscopic Myotomy
Acronym: POEM
Status: Completed | Type: Observational
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Santiago Horgan, Professor of Surgery, University of California, San Diego
Other Study IDs: 091170, 150261
Record Dates: First submitted 2011-07-21; First posted 2011-07-26 (Estimated); Last update posted 2020-03-10 (Actual); Status verified 2018-04

CONDITIONS: Achalasia
Keywords: achalasia; myotomy; endoscopic myotomy; difficulty swallowing
MeSH Terms: conditions — Esophageal Achalasia; Deglutition Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Per-oral endoscopic myotomy
  Interventions: Procedure: Per-oral enodscopic myotomy

INTERVENTIONS:
Procedure: Per-oral enodscopic myotomy
  Other Names: POEM

SUMMARY:
This is a prospective chart review/data collection study of the per oral endoscopic myotomy (POEM) procedure, that will include questionnaires administered throughout the study. Subjects enrolled will be those intending to have a POEM procedure. Data will be collected and reviewed through 12 months post-op.

ELIGIBILITY:
Inclusion:

1. Diagnosis of achalasia
2. Age 18-75
3. Mentally competent to give informed consent
4. Scheduled to undergo a POEM procedure

Exclusion:

1. Pregnant women
2. Any prior surgical treatment for achalasia

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients between the ages of 18-75 who present in the UC San Diego Surgical Specialties clinic with the diagnosis of achalasia will be offered participation in this study.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2009-11; Primary Completion 2019-11 (Actual); Study Completion 2019-11 (Actual)

PRIMARY OUTCOMES:
To evaluate the outcomes of the per-oral endoscopic myotomy (POEM) procedure for the treatment of achalasia | 1 year

SECONDARY OUTCOMES:
To assess the quality of life, pain, and complications of the POEM approach | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Santiago Horgan, M.D., FACS, Principal Investigator — UCSD
Locations (1):
- University of California, San Diego, San Diego, California, United States